CLINICAL TRIAL: NCT00952874
Title: Microsatellite Instability in Anal Squamous Cell Carcinomas of HIV-Positive Versus HIV-Negative Patients
Brief Title: Molecular Biology of Anal Cancer in HIV-Positive Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Lausanne Hospitals (Other); University of Zurich (Other)
Responsible Party: Pascal Gervaz, Department of Surgery, University Hospital Geneva
Other Study IDs: SCCA/HIV
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2009-08

CONDITIONS: Carcinoma; HIV Infections
Keywords: anal cancer; Molecular biology; HIV status; HPV infection; Microsatellite instability; Biopsy proven Squamous Cell carcinoma of the Anus; Squamous Cell carcinoma of the Anus
MeSH Terms: conditions — Carcinoma; HIV Infections; Anus Neoplasms; Papillomavirus Infections; Microsatellite Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biosie of anal cancer
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The molecular mechanisms involved in squamous cell carcinoma of the anus (SCCA) are poorly elucidated. HIV-positive and renal transplant patients are at high risk for developing SCCA, indicating that immune suppression plays a facilitating role. The investigators previously demonstrated that chromosomal instability (CIN) was more prevalent in SCCA of HIV-negative than HIV-positive patients. Hence, the investigators postulate that microsatellite instability (MSI), another molecular pathway, might be a feature of SCCA progression in the HIV-positive population.

Study Aims:

1. to determine the prevalence of MSI in paraffin-embedded tumor specimen of 15 patients from the Swiss HIV cohort who underwent surgical excision for SCCA; and
2. eventually, to test our hypothesis by assessing the MSI status of SCCA in 15 recently operated HIV-negative patients.

Study Design:

The study is designed in two steps:

1. Firstly, the investigators will retrieve tumor specimen from 15 HIV-positive patients, with a biopsy-confirmed diagnosis of SCCA, in three institutions. DNA from tumor and normal tissues will be extracted, and then amplified by PCR. Presence of MSI in tumors will be determined by assessing the microsatellite markers BAT25, BAT26, and CAT25.
2. Secondly, the results of molecular analysis will be compared with a population of HIV-negative patients, with the same tumors, using the same detection technique for MSI.

DETAILED DESCRIPTION:
Background:

In the highly active antiretroviral therapy (HAART) era, the incidence of many cancers remains higher in the HIV-positive than in the general population. This is not only true for AIDS-defining malignancies, such as Kaposi's sarcoma or lymphoma, but also for other cancers, which comprise 58% of all neoplasms in a recently described US cohort [1]. This trend has generated renewed interest in understanding the molecular mechanisms of carcinogenesis in the immune suppressed patient. Potential explanations include prolonged survival of patients with HIV on HAART, high incidence of co-infection with oncogenic viruses, and exposure to risks such as smoking and alcohol [2].

Squamous cell carcinoma of the anus (SCCA) requires integration of human papillomavirus (HPV) DNA into anal canal cell chromosomes. HIV-positive men are at increased risk for developing anal cancer. A Swiss study linking the Swiss HIV cohort study and Swiss cantonal cancer registries has shown greatly elevated SIRs for anal cancer (SIR = 33.4, 95% CI = 10.5-78.6) [3]. Clearly, HPV-HIV coinfection plays a major role in SCCA development, but whether this contribution is associated with distinct molecular pathway of carcinogenesis, remains hypothetical [4].

Anal cancer occurs earlier in HIV-positive individuals (mean age 37 years) compared with HIV-negative men (58 years) and HIV-negative women (65 years). This difference of two decades in age of onset supports the hypothesis that the biology of SCCA differs between HIV-positive and HIV-negative patients [5]. The effect of HIV infection on the natural history of anal HPV infection is poorly understood, but most experts agree on two points: 1) 95% of HIV-positive homosexual men are co-infected with HPV; and 2) HIV infection favors persistence of HPV infection within the ano-genital tract (uterine cervix, vagina, and anal canal).

Two major and mutually exclusive types of genomic instability are involved in cancer progression. The first, known as chromosomal instability (CIN), results from a series of genetic changes, including activation of oncogenes and inactivation of tumor-suppressor genes such as p53 and APC. The second, known as microsatellite instability (MSI), results from somatic (acquired) inactivation of DNA mismatch repair genes (MMR), such as MLH1 (by hypermethylation of its promoter), typically leading to mutation of genes with coding microsatellites, such as BAT 25, BAT26 and CAT25, transforming growth factor receptor II (TGF-RII) and BAX [6].

MSI reflects genomewide instability (resulting from a deficient MMR system), and occurs at increased frequency in HIV-associated cervical intraepithelial and lung neoplasia. In both cases, the frequency of MSI was six fold greater in the HIV-associated tumors, compared with tumors of HIV-indeterminate patients [7]. Others authors have also reported a high rate of MSI in Kaposi's sarcomas and aggressive lymphomas obtained from HIV-infected patients, whereas there is no evidence of similar instability in lesions from HIV-negative patients [8]. The recent observation that the MSI phenotype is restricted to HIV-related lymphomas suggests that a cardinal feature of cancer, such as genetic instability, can be highly influenced by host immunity [9].

MSI status of SCCA in HIV-positive patients has never been investigated, but we have performed a CIN analysis of tumor specimens from 18 HIV- and 10 HIV+ patients diagnosed with SCCA in two US institutions [10]. Tumors in HIV-negative patients were more likely to present CIN than were tumors in HIV-positive patients (24.1% versus 6.6%, P<0.001). Consistent loss of heterozygosity (LOH) on chromosomes 17p, 18q, 5q, and 11q was observed in HIV-negative patients with SCCA. By contrast, allelic loss at 17p, 5q, and 18q was virtually absent in tumors of HIV-positive individuals, indicating that immune suppression promote SCCA progression through an alternate pathway to CIN.

Own Research in the Field:

The applicant is a colorectal surgeon, directly involved in the treatment of patients with anorectal malignancies since 2001. He has collected preliminary data showing specific patterns of molecular aberrations in HIV-related SCCA. These findings have been published in peer-reviewed journals, with the consequence that the applicant is regularly solicited by Editors to write expert opinions and state of the art reviews in the field.

The Swiss cohort of HIV-positive patients will provide a unique opportunity to conduct this research, because of the large number of individuals already enrolled in the existing database, and the existing expertise in the field developed by Professor Hirschel and his team. A large population of patients is indeed a sine qua none condition to start this project due to the relative rarity of these tumors.

Last but not least, the molecular aspect of this research will be conducted in the laboratory of Dr Pierre Hutter, PhD, who is a leader in our country for the detection of hereditary non-polyposis colorectal cancer (HNPCC). Thus, Dr Hutter laboratory will provide an excellent environment to perform the molecular analyses described herein.

Study Hypotheses:

We hypothesize that, in the HIV population, microsatellite instability, rather than chromosomal instability, is the favoured pathway for rapid progression of anal intra-epithelial neoplasia towards invasive SCCA. The second hypothesis is that, by comparison, MSI is either absent or at least very rare in SCCA of HIV-negative individuals.

Study Aims and Objectives

The primary objective of this study is to assess microsatellite instability status in tumor specimens of 15 HIV-positive patients from the Swiss Cohort who were diagnosed with SCCA; an interim analysis will then be performed to determine the incidence of MSI in SCCA of HIV-positive patients. If a majority of tumours exhibit MSI in this population, we will proceed with the second part of the study, which objective is to perform the same analyses in similar tumors of 15 HIV-negative patients, and thus to compare the molecular profiles of SCCA in both populations. By doing so, the potential role of immune suppression in carcinogenesis progression might be established.

Study Design and Plan

Patients:

Patients from the Swiss HIV cohort with a biopsy-proven diagnosis of squamous cell carcinoma of the anus will be identified using the existing database. We choose to analyse at least 15 samples, depending on availability, between 3 SHCS centers. Tumors from HIV-negative patients who underwent surgery for SCCA will be retrieved from the Department of Pathology of University Hospital Geneva, pending review of the protocol by the local Ethics Committee.

Intervention:

All tumor samples will be reassessed for confirmation of diagnosis by a pathologist. For each patient, paraffin blocks with both tumor tissue and normal mucosa will be selected for DNA extraction and polymerase chain reaction at microsatellite targets. The tissues were routinely collected from the operating room, fixed in buffered formalin, embedded in paraffin, and stored for a variable number of months prior to selection for analysis. Paraffin-embedded blocks will be cut with a microtome into 20-µm thick sections. Using a sterile scalpel blade, areas of normal (non-tumor) and cancer tissue will be microdissected under a dissecting microscope utilizing a haematoxylin and eosin-stained section as a guide. The specimens will be deparaffinised in toluol, purified with absolute ethanol, and centrifuged at 14,000 rpm. Previous experience in Dr Hutter's laboratory has demonstrated that it is indeed technically possible to perform this type of molecular analysis in paraffin-embedded tumour specimen.

We will use the reference panel of microsatellite primers recommended for colorectal cancer specimens to determine the presence of microsatellite instability in SCCA. These include the microsatellite markers BAT25, BAT26, as well as CAT25.

Study Evaluations:

Initial evaluation of data will be performed after analysis of the first 15 tumours specimen. If MSI is detected in the HIV-positive population, further investigation will be conducted in tumors of HIV-negative patients. Data analysis will be subject to progress reports conducted with all investigators at regular intervals. We chose to restrict, at least initially, our analysis to 15 tumours for three reasons:

1. This is a relatively rare cancer, and it is unlikely that we will be able to retrieve more than 25 SCCA patients from the Swiss HIV cohort.
2. Our previous study was conducted with 18 tumours specimen in each group, and the differences between groups were statistically significant.
3. This is a pilot exploratory study, and the working hypothesis may prove wrong; it is therefore critical to limit the initial costs in accordance with the study budget and availability of Dr Hutter's expertise. If our hypothesis is supported by the initial results, we may proceed with additional investigations and a more elaborated research project with adequate funding resources.¨ For these reasons, we will restrict our research to three SHCS centers. Zurich, Geneva and Lausanne were chosen essentially based on existing relationship between the visceral surgery units.

Data Analysis:

MSI status of tumors will be assessed by Pierre Hutter. The results will then be correlated with the epidemiological data from the Swiss cohort, and correlated with the patients' clinical characteristics, including viral load, CD4+ count, as well as clinical outcome. The results will also be correlated with treatment outcome and cancer survival.

Time Frame:

Tumor specimen will be retrieved from the Departments of Pathology in Lausanne, Geneva and Zurich in the beginning of 2009. The MSI analysis is a straightforward procedure, which takes about 24 hours in the laboratory of Dr Hutter. Thus, the analysis of the 15 specimen in the HIV-positive population will be completed by the end of March 2009. Further decision regarding subsequent analyses in the HIV-negative population will then be subjected to decision, according to the results obtained in these initial tumors.

Status of Ethical Approval:

Patients enrolled in the Swiss HIV cohort study initially gave their consent for participating in this type of study. Almost all patients at the HIV centres consented to take part in genetic research in order to identify specific factors that might result in differences in the course of the disease. Obviously, all analyses will be performed on tumor specimen, and these will not be traceable to the patients' identities. Thus, all genetic testing will be totally anonymous. By contrast, further approval by the local Ethics Committee in Geneva will be sought, should the analysis be performed on tumor specimen from HIV-negative patients.

Study budget:

The initial analysis of 15 HIV-positive patients will be performed free of charge by Pierre Hutter. The cost for molecular study is estimated at 250.-CHF per case. Thus, in case the analysis of MSI in this group leads to promising results, it is estimated that the cost of analysis in 12-15 HIV-negative patients will cost around 3,000.-CHF. Funding for this type of research will be available through the Fonds de Service of Department of Surgery at University Hospital Geneva.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven Squamous cell carcinoma of the anus
* Informed consent

Exclusion Criteria:

* None

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive and negative patients with biopsy proven squamous cell carcinoma of the anal canal
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Hirschel, Study Chair — Swidd HIV cohort
Locations (1):
- University Hospital Geneva, Geneva, Switzerland